CLINICAL TRIAL: NCT00473083
Title: A Randomized Controlled Trial of Systemic and Topical Treatments for Rash Secondary to Erlotinib in Advanced Stage IIIB or IV Non-Small Cell Lung Cancer
Brief Title: Systemic and Topical Treatments for Rash Secondary to Erlotinib in Lung Cancer
Acronym: LUTRAERL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML21016
Record Dates: First submitted 2007-05-10; First posted 2007-05-14 (Estimated); Results first posted 2017-04-04 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2017-02

CONDITIONS: Rash
Keywords: Rash; Erlotinib; Lung Cancer
MeSH Terms: conditions — Exanthema; Lung Neoplasms | interventions — Minocycline; Clindamycin; Hydrocortisone; Erlotinib Hydrochloride; Triamcinolone Acetonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1: Prophylactic Treatment (Experimental): Participants will receive prophylactic treatment with minocycline 100 mg orally twice-daily for at least 4 weeks on the initiation of erlotinib therapy. If rash occurs during the 4 week period of minocycline prophylaxis, the minocycline prophylaxis will continue and additional treatment by grade of rash will be according to the Treatment Arm 2 schedule. If rash occurs after the completion of the 4 week prophylaxis period, treatment by grade of rash will be according to the Treatment Arm 2 schedule.
  Interventions: Drug: Minocycline; Drug: Clindamycin 2% in hydrocortisone 1% lotion; Drug: Erlotinib; Drug: Topical clindamycin 2%, triamcinolone acetonide 0.1% soln
- Arm 2: Reactive Treatment (Experimental): Pts will receive treatment at initiation of rash. Tx is dependent on grading of rash as follows:
  Grade 1 or 2A: Topical clindamycin 2%, with hydrocortisone 1% in lotion base applied twice daily until resolution of rash by one grade
  Grade 2B: Topical clindamycin 2%, with hydrocortisone 1% in lotion base applied 2x daily and oral minocycline 100mg 2x daily for a min. of 4 weeks and continuing thereafter, as required, until resolution of rash by 1 grade. Scalp lesions will be treated with a topical clindamycin 2%, triamcinolone acetonide 0.1% soln.
  Grade 3: Pts will discontinue tx with erlotinib 150mg for 1 week and restart at 100mg once daily.
  Tx with topical clindamycin 2%, with hydrocortisone 1% in lotion base applied 2x daily and oral minocycline 100mg 2x daily for a min. of 4 weeks and continuing thereafter, as required, until resolution of rash to Grade 1 or 2A. Scalp lesions will be treated with a topical clindamycin 2%, triamcinolone acetonide 0.1% soln.
  Interventions: Drug: Minocycline; Drug: Clindamycin 2% in hydrocortisone 1% lotion; Drug: Erlotinib; Drug: Topical clindamycin 2%, triamcinolone acetonide 0.1% soln
- Arm 3: No Treatment Unless Severe (Grade 3) (Experimental): This is the control group. Patients will be treated only if grade 3 rash develops. For grade 3 rash, treatment will be in accordance with that of Grade 3 rash in Treatment Arm 2.
  Interventions: Drug: Minocycline; Drug: Clindamycin 2% in hydrocortisone 1% lotion; Drug: Erlotinib; Drug: Topical clindamycin 2%, triamcinolone acetonide 0.1% soln

INTERVENTIONS:
Drug: Minocycline — Patients will receive prophylactic treatment with minocycline 100 mg orally twice-daily for at least 4 weeks on the initiation of erlotinib therapy. If rash occurs during the 4 week period of minocycline prophylaxis, the minocycline prophylaxis will continue and additional treatment by grade of rash will be according to the Treatment Arm 2 schedule. If rash occurs after the completion of the 4 week prophylaxis period, treatment by grade of rash will be according to the Treatment Arm 2 schedule.
  Other Names: Dynacin; Minocin; Minocin PAC; Solodyn; Vectrin; Myrac
Drug: Clindamycin 2% in hydrocortisone 1% lotion — Appropriate amounts of clindamycin and hydrocortisone powder are mixed with corresponding amount of Nutraderm® lotion for this mixture.
  If preferred, the appropriate amount of clindamycin powder can be mixed with Emo-Cort® lotion (already contains hydrocortisone 1%), available in 60 mL bottles.
Drug: Erlotinib — Erlotinib will be given on an outpatient basis at a fixed dose of either 150 or 100 mg as a single daily oral dose.
  Other Names: Tarceva
Drug: Topical clindamycin 2%, triamcinolone acetonide 0.1% soln — Clindamycin 2% in Triamcinolone acetonide 0.1% solution in equal parts propylene glycol and water

SUMMARY:
The purpose of this trial is to determine if rash caused by erlotinib can be successfully treated and if so to determine the optimal treatment approach.

Hypothesis:

Hypothesis 1: If the incidence of rash is 50% while on erlotinib, prophylactic monotherapy with minocycline can prevent occurrence in 50% of these patients.

Hypothesis 2: Treatment of rash is successful in improving rash by at least one Grade in 80% of patients.

Hypothesis 3: In patients with untreated rash, the rash will be self-limiting in 25% of patients, and 65% will be grade 1, 2A, and 2b. Ten percent will be grade 3 requiring treatment with monotherapy intervention.

DETAILED DESCRIPTION:
Erlotinib has been shown to prolong survival in NSCLC patients who are no longer candidates for further chemotherapy. In July 2005, erlotinib was approved in Canada for the treatment of patients with locally advanced or metastatic NSCLC, following failure of first or second-line chemotherapy.

Erlotinib's side effect profile includes rash. The incidence of rash in clinical trials has been reported to be approximately 50 - 75%, and has been hypothesised to parallel tumour response (20).

The treatment of rash is controversial and many oncologists believe it is untreatable and self-limiting. The cause of the rash is not well understood but is felt to be a systemic event. Clinical experience of the investigators has suggested that minocycline 100 mg orally given twice-daily for 4 weeks and clindamycin 2% and hydrocortisone 1% topical cream for moderate to severe rash is a successful treatment.

The objectives of this trial are to better delineate the rash and its features and to describe an optimal treatment. Since the rash is often facial in distribution and can therefore lead to physical and psychological distress to the patient, a dermatology life quality index will also be completed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytological documented diagnosis of inoperable, locally advanced, recurrent or metastatic (stage IIIB or stage IV) non-small cell lung cancer.
2. Evidence of disease (measurable disease is not mandatory).
3. 18 years of age or older.
4. ECOG performance status of 0 - 3.
5. Written informed consent prior to study-specific screening procedures, with the understanding that the patient has the right to withdraw from the study at any time, without prejudice.

Exclusion Criteria:

1. A history of another cancer other than basal cell carcinoma or cervical cancer in situ within the past 3 years
2. Prior therapy with any type of cancer growth factor inhibitor (EGFR inhibitor or agent targeting this family of growth factor receptors)
3. Life expectancy of less than 12 weeks.
4. Ongoing toxic effects from prior chemotherapy.
5. Pregnant or lactating women.
6. Females of childbearing potential who have a positive or no pregnancy test (pregnancy tests must be obtained within 72 hours before starting therapy). (Postmenopausal women must have been amenorrheic for at least 12 months to be considered of non-childbearing potential).
7. Male or female patients with reproductive potential who are unwilling to use effective and reliable contraceptive methods throughout the course of the study and for 90 days after the last dose of study medication.
8. Ongoing treatment with any inhibitors or inducers of CYP3A4 activity
9. Any unstable systemic disease (including active infection, grade 4 hypertension, unstable angina, congestive heart failure, hepatic, renal or metabolic disease).
10. Any significant ophthalmologic abnormality, especially severe dry eye syndrome, keratoconjunctivitis sicca, Sjögren syndrome, severe exposure keratitis or any other disorder likely to increase the risk of corneal epithelial lesions.
11. Unwilling or unable to comply with the protocol for the duration of the study.
12. Patients who have experienced prior hypersensitivity reaction to active ingredients or excipients of the following compounds: erlotinib, minocycline, tetracycline, doxycycline or clindamycin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2009-01; Primary Completion 2012-12 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barb Melosky, MD, Principal Investigator — British Columbia Cancer Agency
Locations (9):
- Canada (9):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - BC Cancer Agency - Abbotsford, Abbotsford, British Columbia
  - Burnaby Hospital Regional Cancer Centre, Burnaby, British Columbia
  - BC Cancer Agency - Fraser Valley Centre, Vancouver, British Columbia
  - BC Cancer Agency Vancouver Centre, Vancouver, British Columbia
  - BC Cancer Agency - Vancouver Island Centre, Victoria, British Columbia
  - Mount Sinai Hospital, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario

REFERENCES:
- [Background] Modjtahedi H, Dean C. The receptor for EGF and its ligands - expression, prognostic value and target for therapy in cancer (review). Int J Oncol. 1994 Feb;4(2):277-96. doi: 10.3892/ijo.4.2.277. PMID 21566922
- [Background] Salomon DS, Brandt R, Ciardiello F, Normanno N. Epidermal growth factor-related peptides and their receptors in human malignancies. Crit Rev Oncol Hematol. 1995 Jul;19(3):183-232. doi: 10.1016/1040-8428(94)00144-i. No abstract available. PMID 7612182
- [Background] Rusch V, Mendelsohn J, Dmitrovsky E. The epidermal growth factor receptor and its ligands as therapeutic targets in human tumors. Cytokine Growth Factor Rev. 1996 Aug;7(2):133-41. doi: 10.1016/1359-6101(96)00016-0. PMID 8899291
- [Background] Davies DE, Chamberlin SG. Targeting the epidermal growth factor receptor for therapy of carcinomas. Biochem Pharmacol. 1996 May 3;51(9):1101-10. doi: 10.1016/0006-2952(95)02232-5. PMID 8645330
- [Background] Veale D, Ashcroft T, Marsh C, Gibson GJ, Harris AL. Epidermal growth factor receptors in non-small cell lung cancer. Br J Cancer. 1987 May;55(5):513-6. doi: 10.1038/bjc.1987.104. PMID 3038157
- [Background] Sekine I, Takami S, Guang SG, Yokose T, Kodama T, Nishiwaki Y, Kinoshita M, Matsumoto H, Ogura T, Nagai K. Role of epidermal growth factor receptor overexpression, K-ras point mutation and c-myc amplification in the carcinogenesis of non-small cell lung cancer. Oncol Rep. 1998 Mar-Apr;5(2):351-4. PMID 9468555
- [Background] Pfeiffer P, Clausen PP, Andersen K, Rose C. Lack of prognostic significance of epidermal growth factor receptor and the oncoprotein p185HER-2 in patients with systemically untreated non-small-cell lung cancer: an immunohistochemical study on cryosections. Br J Cancer. 1996 Jul;74(1):86-91. doi: 10.1038/bjc.1996.320. PMID 8679464
- [Background] Cerny T, Barnes DM, Hasleton P, Barber PV, Healy K, Gullick W, Thatcher N. Expression of epidermal growth factor receptor (EGF-R) in human lung tumours. Br J Cancer. 1986 Aug;54(2):265-9. doi: 10.1038/bjc.1986.172. PMID 3017396
- [Background] IMPATH Inc. Analysis of EGFr Expression in a selection of tumour types. IMPATH Study Number PFZ04. 1998-1999:1-16.
- [Background] Reissmann PT, Koga H, Figlin RA, Holmes EC, Slamon DJ. Amplification and overexpression of the cyclin D1 and epidermal growth factor receptor genes in non-small-cell lung cancer. Lung Cancer Study Group. J Cancer Res Clin Oncol. 1999;125(2):61-70. doi: 10.1007/s004320050243. PMID 10190311
- [Background] Fujino S, Enokibori T, Tezuka N, Asada Y, Inoue S, Kato H, Mori A. A comparison of epidermal growth factor receptor levels and other prognostic parameters in non-small cell lung cancer. Eur J Cancer. 1996 Nov;32A(12):2070-4. doi: 10.1016/s0959-8049(96)00243-2. PMID 9014747
- [Background] Fontanini G, Vignati S, Bigini D, Mussi A, Lucchi H, Angeletti CA, Pingitore R, Pepe S, Basolo F, Bevilacqua G. Epidermal growth factor receptor (EGFr) expression in non-small cell lung carcinomas correlates with metastatic involvement of hilar and mediastinal lymph nodes in the squamous subtype. Eur J Cancer. 1995;31A(2):178-83. doi: 10.1016/0959-8049(93)00421-m. PMID 7718322
- [Background] Rusch V, Klimstra D, Venkatraman E, Pisters PW, Langenfeld J, Dmitrovsky E. Overexpression of the epidermal growth factor receptor and its ligand transforming growth factor alpha is frequent in resectable non-small cell lung cancer but does not predict tumor progression. Clin Cancer Res. 1997 Apr;3(4):515-22. PMID 9815714
- [Background] Ohsaki Y, Toyoshima E, Fujiuchi S, Nishigaki Y, Kikuchi K. EGR receptor (EGFR) expression correlates poor prognosis in non-small cell lung cancer (NSCLC) patients interacting with p53 overexpression (abstract). Proc Am Assoc Cancer Res 1997; 38:327.
- [Background] Lei W, Mayotte JE, Levitt ML. Enhancement of chemosensitivity and programmed cell death by tyrosine kinase inhibitors correlates with EGFR expression in non-small cell lung cancer cells. Anticancer Res. 1999 Jan-Feb;19(1A):221-8. PMID 10226546
- [Background] Veale D, Kerr N, Gibson GJ, Kelly PJ, Harris AL. The relationship of quantitative epidermal growth factor receptor expression in non-small cell lung cancer to long term survival. Br J Cancer. 1993 Jul;68(1):162-5. doi: 10.1038/bjc.1993.306. PMID 8391303
- [Background] Busam KJ, Capodieci P, Motzer R, Kiehn T, Phelan D, Halpern AC. Cutaneous side-effects in cancer patients treated with the antiepidermal growth factor receptor antibody C225. Br J Dermatol. 2001 Jun;144(6):1169-76. doi: 10.1046/j.1365-2133.2001.04226.x. PMID 11422037
- [Background] Van Doorn R, Kirtschig G, Scheffer E, Stoof TJ, Giaccone G. Follicular and epidermal alterations in patients treated with ZD1839 (Iressa), an inhibitor of the epidermal growth factor receptor. Br J Dermatol. 2002 Sep;147(3):598-601. doi: 10.1046/j.1365-2133.2002.04864.x. PMID 12207609
- [Background] Herbst RS, LoRusso PM, Purdom M, Ward D. Dermatologic side effects associated with gefitinib therapy: clinical experience and management. Clin Lung Cancer. 2003 May;4(6):366-9. doi: 10.3816/clc.2003.n.016. PMID 14599302
- [Background] Perez-Soler R, Saltz L. Cutaneous adverse effects with HER1/EGFR-targeted agents: is there a silver lining? J Clin Oncol. 2005 Aug 1;23(22):5235-46. doi: 10.1200/JCO.2005.00.6916. PMID 16051966
- [Background] Shepherd FA, Rodrigues Pereira J, Ciuleanu T, Tan EH, Hirsh V, Thongprasert S, Campos D, Maoleekoonpiroj S, Smylie M, Martins R, van Kooten M, Dediu M, Findlay B, Tu D, Johnston D, Bezjak A, Clark G, Santabarbara P, Seymour L; National Cancer Institute of Canada Clinical Trials Group. Erlotinib in previously treated non-small-cell lung cancer. N Engl J Med. 2005 Jul 14;353(2):123-32. doi: 10.1056/NEJMoa050753. PMID 16014882
- [Background] Perez-Soler R, Delord JP, Halpern A, Kelly K, Krueger J, Sureda BM, von Pawel J, Temel J, Siena S, Soulieres D, Saltz L, Leyden J. HER1/EGFR inhibitor-associated rash: future directions for management and investigation outcomes from the HER1/EGFR inhibitor rash management forum. Oncologist. 2005 May;10(5):345-56. doi: 10.1634/theoncologist.10-5-345. PMID 15851793
- [Result] Melosky B, Anderson H, Burkes RL, Chu Q, Hao D, Ho V, Ho C, Lam W, Lee CW, Leighl NB, Murray N, Sun S, Winston R, Laskin JJ. Pan Canadian Rash Trial: A Randomized Phase III Trial Evaluating the Impact of a Prophylactic Skin Treatment Regimen on Epidermal Growth Factor Receptor-Tyrosine Kinase Inhibitor-Induced Skin Toxicities in Patients With Metastatic Lung Cancer. J Clin Oncol. 2016 Mar 10;34(8):810-5. doi: 10.1200/JCO.2015.62.3918. Epub 2015 Nov 16. PMID 26573073

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible patients had a histological or cytologic documented diagnosis of metastatic NSCLC, with and Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 3. The study was initiated on November 7, 2008, and concluded with the last patient in December 2012.
Groups:
- Arm 1: Prophylactic Treatment: Subjects (approximately 50) will be given minocycline (an antibiotic pill) 100mg orally to take for 4 weeks at the same time as starting their erlotinib to see if the rash can be prevented
  minocycline: Arm 1: Subjects (approximately 50) will be given minocycline (an antibiotic pill) 100mg orally to take for 4 weeks at the same time as starting their erlotinib to see if the rash can be prevented. If rash occurs then subjects will be treated using a medicated lotion, (clindamycin 2% and hydrocortisone 1%,) to be applied to the rash and if the rash is more severe, minocycline may be continued for more than 4 weeks.
- Arm 2: Reactive Treatment: Arm 2: Subjects (Approximately 50) will be treated for the rash caused by erlotinib when it develops and the treatment will be a medicated lotion, (clindamycin 2% and hydrocortisone 1%,), applied to the rash and if the rash is more severe, minocycline 100mg orally twice daily. Scalp lesions will be treated with a topical clindamycin 2 %, triamcinolone acetonide 0.1% solution.
  minocycline; Lotion (clindamycin 2% /hydrocortisone 1%): Subjects (Approximately 50) will be treated for the rash caused by erlotinib when it develops and the treatment will be a medicated lotion, (clindamycin 2% and hydrocortisone 1%,), applied to the rash and if the rash is more severe, minocycline 100mg orally twice daily. Scalp lesions will be treated with a topical clindamycin 2 %, triamcinolone acetonide 0.1% solution
- Arm 3: No Treatment Unless Severe (Grade 3): Arm 3: Subjects (Approximately 50) that develop the rash caused by erlotinib will only be treated if their rash becomes severe to see if it will go away itself. The treatment for severe rash will be medicated lotion, (clindamycin 2% and hydrocortisone 1%,), applied to the rash and minocycline 100mg orally twice daily. Scalp lesions will be treated with a topical clindamycin 2 %, triamcinolone acetonide 0.1% solution
  clindamycin 2% and hydrocortisone 1%,: Arm 3: Subjects (Approximately 50) that develop the rash caused by erlotinib will only be treated if their rash becomes severe to see if it will go away itself. The treatment for severe rash will be medicated lotion, (clindamycin 2% and hydrocortisone 1%,), applied to the rash and minocycline 100mg orally twice daily. Scalp lesions will be treated with a topical clindamycin 2 %, triamcinolone acetonide 0.1% solution.
Period: Overall Study
Arm/Group | Arm 1: Prophylactic Treatment | Arm 2: Reactive Treatment | Arm 3: No Treatment Unless Severe (Grade 3)
Started | 50 | 50 | 50
Completed | 49 (One patient (2%) from treatment arm 1 discontinued the study drug as a result of a TEAE (dizziness)) | 50 | 50
Not Completed | 1 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm 2: Reactive Treatmen: Arm 2: Subjects (Approximately 50) will be treated for the rash caused by erlotinib when it develops and the treatment will be a medicated lotion, (clindamycin 2% and hydrocortisone 1%,), applied to the rash and if the rash is more severe, minocycline 100mg orally twice daily. Scalp lesions will be treated with a topical clindamycin 2 %, triamcinolone acetonide 0.1% solution.
  minocycline; Lotion (clindamycin 2% /hydrocortisone 1%): Subjects (Approximately 50) will be treated for the rash caused by erlotinib when it develops and the treatment will be a medicated lotion, (clindamycin 2% and hydrocortisone 1%,), applied to the rash and if the rash is more severe, minocycline 100mg orally twice daily. Scalp lesions will be treated with a topical clindamycin 2 %, triamcinolone acetonide 0.1% solution
- Total: Total of all reporting groups
Arm/Group | Arm 1: Prophylactic Treatment | Arm 2: Reactive Treatmen | Arm 3: No Treatment Unless Severe (Grade 3) | Total
Number analyzed (Participants) | 50 | 50 | 50 | 150
Age, Continuous [Median (Full Range); unit: years] | 64.3 [30 to 79] | 65.9 [48 to 83] | 64.4 [46 to 82] | 64.9 [30 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 27 | 27 | 71
  Male | 33 | 23 | 23 | 79
Region of Enrollment [Number; unit: participants]
  Canada | 50 | 50 | 50 | 150

OUTCOME MEASURES:

1. Primary Outcome: Overall Incidence of Rash
Description: The overall incidence of any grade of erlotinib-induced rash among the three treatment arms.
  For overall incidence of rash a binary variable will be designed. Data will be summarized with percentages by treatment group.
Time Frame: From onset of rash until resolution, up to 4 weeks following progression, an average of 1 year
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1: Prophylactic Treatment | Arm 2: Reactive Treatment | Arm 3: No Treatment Unless Severe (Grade 3)
Number analyzed (Participants) | 50 | 50 | 50
percentage of participants | 84 | 84 | 82
Statistical Analysis 1: Comparison: Arm 1: Prophylactic Treatment vs Arm 2: Reactive Treatment vs Arm 3: No Treatment Unless Severe (Grade 3); Test type: Superiority or Other; p = 0.8769, Chi-squared — P for arm 1 v arms 2 and 3 combined
Statistical Analysis 2: Comparison: Arm 1: Prophylactic Treatment vs Arm 2: Reactive Treatment vs Arm 3: No Treatment Unless Severe (Grade 3); Test type: Superiority or Other; p = 0.147, Wilcoxon (Mann-Whitney) — P for arm 1 v arms 2 and 3 combined

2. Primary Outcome: Time Duration From Onset of Rash Until Resolution
Description: To investigate if the rash caused by erlotinib is self-limiting.
  A time variable will be defined to identify the duration from onset of rash until resolution. Resolution will be defined as resolution to severity Grade 1 for patients with rash of maximum severity grade >1 and resolution to Grade 0 for patients with maximum rash severity = 1. For patients where resolution is not observed the time considered will be the maximum time from onset of rash until end of the study.
  The analyses will be performed using the following two sub-populations: subjects with maximum severity of rash of Grade 1, 2a and 2b will constitute one sub-population and Grade 3 will be considered the second sub-population.
  The comparisons will be performed primarily for Group 1 vs. Group 3 and Group 2 vs. Group 3 and secondly for Group 1 vs. Group 2.
Time Frame: From onset of rash until resolution, up to 4 weeks following progression, an average of 1 year
Population: Patients With Maximum Severity of Rash Grade 1, 2b: Arm 1 (n=36), Arm 2 (n=38), Arm 3 (n=27)
  Patients With Maximum Severity of Rash Grade 3: Arm 1 (n=6), Arm 2 (n=4), Arm 3 (n=14)
Measure: Median (Inter-Quartile Range); unit: days
Groups:
- Arm 1: Prophylactic Treatment: Subjects will be given minocycline (an antibiotic pill) 100mg orally to take for 4 weeks at the same time as starting their erlotinib to see if the rash can be prevented
  minocycline: Arm 1: Subjects will be given minocycline (an antibiotic pill) 100mg orally to take for 4 weeks at the same time as starting their erlotinib to see if the rash can be prevented. If rash occurs then subjects will be treated using a medicated lotion, (clindamycin 2% and hydrocortisone 1%,) to be applied to the rash and if the rash is more severe, minocycline may be continued for more than 4 weeks.
- Arm 2: Reactive Treatment: Arm 2: Subjects will be treated for the rash caused by erlotinib when it develops and the treatment will be a medicated lotion, (clindamycin 2% and hydrocortisone 1%,), applied to the rash and if the rash is more severe, minocycline 100mg orally twice daily. Scalp lesions will be treated with a topical clindamycin 2 %, triamcinolone acetonide 0.1% solution.
  minocycline; Lotion (clindamycin 2% /hydrocortisone 1%): Subjects will be treated for the rash caused by erlotinib when it develops and the treatment will be a medicated lotion, (clindamycin 2% and hydrocortisone 1%,), applied to the rash and if the rash is more severe, minocycline 100mg orally twice daily. Scalp lesions will be treated with a topical clindamycin 2 %, triamcinolone acetonide 0.1% solution
- Arm 3: No Treatment Unless Severe (Grade 3): Arm 3: Subjects that develop the rash caused by erlotinib will only be treated if their rash becomes severe to see if it will go away itself. The treatment for severe rash will be medicated lotion, (clindamycin 2% and hydrocortisone 1%,), applied to the rash and minocycline 100mg orally twice daily. Scalp lesions will be treated with a topical clindamycin 2 %, triamcinolone acetonide 0.1% solution
  clindamycin 2% and hydrocortisone 1%,: Arm 3: Subjects that develop the rash caused by erlotinib will only be treated if their rash becomes severe to see if it will go away itself. The treatment for severe rash will be medicated lotion, (clindamycin 2% and hydrocortisone 1%,), applied to the rash and minocycline 100mg orally twice daily. Scalp lesions will be treated with a topical clindamycin 2 %, triamcinolone acetonide 0.1% solution.
Arm/Group | Arm 1: Prophylactic Treatment | Arm 2: Reactive Treatment | Arm 3: No Treatment Unless Severe (Grade 3)
Number analyzed (Participants) | 42 | 42 | 41
days
  Patients With Max Severity of Rash Gr 1, 2a and 2b: number analyzed (Participants) | 36 | 38 | 27
  Patients With Max Severity of Rash Gr 1, 2a and 2b | 133.0 [80.5 to 308.5] | 92.0 [51.0 to 301.0] | 98.0 [47.0 to 143.0]
  Patients With Maximum Severity of Rash Grade 3: number analyzed (Participants) | 6 | 4 | 14
  Patients With Maximum Severity of Rash Grade 3 | 201.0 [77.0 to 449.0] | 76.0 [56.5 to 90.5] | 54.0 [50.0 to 158.0]
Statistical Analysis 1: Comparison: Arm 1: Prophylactic Treatment vs Arm 2: Reactive Treatment; Test type: Superiority or Other; p = 0.1503, Wilcoxon (Mann-Whitney) — P(arm 1 v arm 2) in patients with maximum severity of rash grade 1, 2a, or 2b
Statistical Analysis 2: Comparison: Arm 2: Reactive Treatment vs Arm 3: No Treatment Unless Severe (Grade 3); Test type: Superiority or Other; p = 0.4681, Wilcoxon (Mann-Whitney) — P(arm2 v arm3) in patients with maximum severity of rash grade 1, 2a, or 2b
Statistical Analysis 3: Comparison: Arm 1: Prophylactic Treatment vs Arm 3: No Treatment Unless Severe (Grade 3); Test type: Superiority or Other; p = 0.0196, Wilcoxon (Mann-Whitney) — P(arm 1 v arm 3) in patients with maximum severity of rash grade 1, 2a, or 2b
Statistical Analysis 4: Comparison: Arm 1: Prophylactic Treatment vs Arm 2: Reactive Treatment; Test type: Superiority or Other; p = 0.1658, Wilcoxon (Mann-Whitney) — P(arm 1 v arm 2) in patients with maximum severity of rash grade 3
Statistical Analysis 5: Comparison: Arm 2: Reactive Treatment vs Arm 3: No Treatment Unless Severe (Grade 3); Test type: Superiority or Other; p > 0.9999, Wilcoxon (Mann-Whitney) — P(arm 2 v arm 3) in patients with maximum severity of rash grade 3. P-value was calculated to be >0.9999 using the Wilcoxon Rank Sumtest by comparing between the two treatment arms
Statistical Analysis 6: Comparison: Arm 1: Prophylactic Treatment vs Arm 3: No Treatment Unless Severe (Grade 3); Test type: Superiority or Other; p = 0.285, Wilcoxon (Mann-Whitney) — P(arm 1 v arm 3) in patients with maximum severity of rash grade 3

3. Secondary Outcome: Severity of Rash Caused by Erlotinib
Description: The maximum severity of rash per subject will be summarized by treatment group. The summary will include only subjects who indicated any occurrence of rash.
Time Frame: Onset until resolution, up to 4 weeks following progression, on average of 1 year
Population: Arm 1 (n=42), Arm 2 (n=42), Arm 3, (n=41)
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1: Prophylactic Treatment | Arm 2: Reactive Treatment | Arm 3: No Treatment Unless Severe (Grade 3)
Number analyzed (Participants) | 42 | 42 | 41
percentage of participants
  Maximal Rash Grade 1 | 40.5 | 47.6 | 46.3
  Maximal Rash Grade 2a | 26.2 | 33.3 | 14.6
  Maximal Rash Grade 2b | 19.0 | 9.5 | 4.9
  Maximal Rash Grade 3 | 14.3 | 9.5 | 34.1
Statistical Analysis 1: Comparison: Arm 1: Prophylactic Treatment vs Arm 2: Reactive Treatment; Maximal Rash Grade 1; Test type: Superiority or Other; p = 0.5097, Chi-squared
Statistical Analysis 2: Comparison: Arm 1: Prophylactic Treatment vs Arm 2: Reactive Treatment; Maximal Rash Grade 2a; Test type: Superiority or Other; p = 0.4740, Chi-squared
Statistical Analysis 3: Comparison: Arm 1: Prophylactic Treatment vs Arm 2: Reactive Treatment; Maximal Severity Grade 2b; Test type: Superiority or Other; p = 0.2123, Chi-squared
Statistical Analysis 4: Comparison: Arm 1: Prophylactic Treatment vs Arm 2: Reactive Treatment; Maximal Severity Grade 3; Test type: Superiority or Other; p = 0.5004, Chi-squared
Statistical Analysis 5: Comparison: Arm 2: Reactive Treatment vs Arm 3: No Treatment Unless Severe (Grade 3); Maximal Severity Grade 1; Test type: Superiority or Other; p = 0.9072, Chi-squared
Statistical Analysis 6: Comparison: Arm 2: Reactive Treatment vs Arm 3: No Treatment Unless Severe (Grade 3); Maximal Severity Grade 2a; Test type: Superiority or Other; p = 0.0464, Chi-squared
Statistical Analysis 7: Comparison: Arm 2: Reactive Treatment vs Arm 3: No Treatment Unless Severe (Grade 3); Maximal Severity Grade 2b; Test type: Superiority or Other; p = 0.6759, Chi-squared
Statistical Analysis 8: Comparison: Arm 2: Reactive Treatment vs Arm 3: No Treatment Unless Severe (Grade 3); Maximal Severity Grade 3; Test type: Superiority or Other; p = 0.0065, Chi-squared
Statistical Analysis 9: Comparison: Arm 1: Prophylactic Treatment vs Arm 3: No Treatment Unless Severe (Grade 3); Maximal Severity Grade 1; Test type: Superiority or Other; p = 0.5898, Chi-squared
Statistical Analysis 10: Comparison: Arm 1: Prophylactic Treatment vs Arm 3: No Treatment Unless Severe (Grade 3); Maximal Severity Grade 2a; Test type: Superiority or Other; p = 0.1921, Chi-squared
Statistical Analysis 11: Comparison: Arm 1: Prophylactic Treatment vs Arm 3: No Treatment Unless Severe (Grade 3); Maximal Severity Grade 2b; Test type: Superiority or Other; p = 0.0882, Chi-squared
Statistical Analysis 12: Comparison: Arm 1: Prophylactic Treatment vs Arm 3: No Treatment Unless Severe (Grade 3); Maximal Severity Grade 3; Test type: Superiority or Other; p = 0.0344, Chi-squared

4. Secondary Outcome: Overall Survival
Time Frame: Until death
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm 1: Prophylactic Treatment | Arm 2: Reactive Treatment | Arm 3: No Treatment Unless Severe (Grade 3)
Number analyzed (Participants) | 50 | 50 | 50
months | 7.6 [4.7 to 12.4] | 8.0 [3.5 to 11.8] | 6.0 [5.5 to 7.3]
Statistical Analysis 1: Comparison: Arm 1: Prophylactic Treatment vs Arm 2: Reactive Treatment vs Arm 3: No Treatment Unless Severe (Grade 3); Test type: Superiority or Other; p = 0.3834, Log Rank

5. Secondary Outcome: Duration of Treatment
Time Frame: Up to one year
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm 1: Prophylactic Treatment | Arm 2: Reactive Treatment | Arm 3: No Treatment Unless Severe (Grade 3)
Number analyzed (Participants) | 50 | 50 | 50
months | 3.6 [2.1 to 4.6] | 1.8 [1.3 to 2.7] | 1.8 [1.7 to 2.4]

6. Secondary Outcome: Time to First Presentation of Rash
Time Frame: Up to onset of rash while on study treatment
Population: Subjects with maximum severity of rash of grade 1, 2a, 2b and 3
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Arm 1: Prophylactic Treatment | Arm 2: Reactive Treatment | Arm 3: No Treatment Unless Severe (Grade 3)
Number analyzed (Participants) | 42 | 42 | 41
days | 17.4 (19.7) | 13.3 (19.0) | 12.0 (11.1)
Statistical Analysis 1: Comparison: Arm 1: Prophylactic Treatment vs Arm 2: Reactive Treatment vs Arm 3: No Treatment Unless Severe (Grade 3); Test type: Superiority or Other; p = 0.0147, Wilcoxon (Mann-Whitney)

7. Primary Outcome: Overall Incidence of Grade 3 Rash
Description: The overall incidence of grade 3 erlotinib-induced rash among the three treatment arms.
  For overall incidence of rash a binary variable will be designed. Data will be summarized with percentages by treatment group.
Time Frame: From onset of rash until resolution, up to 4 weeks following progression, on average of 1 year
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1: Prophylactic Treatment | Arm 2: Reactive Treatment | Arm 3: No Treatment Unless Severe (Grade 3)
Number analyzed (Participants) | 50 | 50 | 50
percentage of participants | 14.3 | 9.5 | 34.1

ADVERSE EVENTS:
Groups:
- Arm 1: Rash Prevention: Subjects (approximately 50) will be given minocycline (an antibiotic pill) 100mg orally to take for 4 weeks at the same time as starting their erlotinib to see if the rash can be prevented
  minocycline: Arm 1: Subjects (approximately 50) will be given minocycline (an antibiotic pill) 100mg orally to take for 4 weeks at the same time as starting their erlotinib to see if the rash can be prevented. If rash occurs then subjects will be treated using a medicated lotion, (clindamycin 2% and hydrocortisone 1%,) to be applied to the rash and if the rash is more severe, minocycline may be continued for more than 4 weeks.
- Arm 2: Treat Only Upon Initiation of Rash: Arm 2: Subjects (Approximately 50) will be treated for the rash caused by erlotinib when it develops and the treatment will be a medicated lotion, (clindamycin 2% and hydrocortisone 1%,), applied to the rash and if the rash is more severe, minocycline 100mg orally twice daily. Scalp lesions will be treated with a topical clindamycin 2 %, triamcinolone acetonide 0.1% solution.
  minocycline; Lotion (clindamycin 2% /hydrocortisone 1%): Subjects (Approximately 50) will be treated for the rash caused by erlotinib when it develops and the treatment will be a medicated lotion, (clindamycin 2% and hydrocortisone 1%,), applied to the rash and if the rash is more severe, minocycline 100mg orally twice daily. Scalp lesions will be treated with a topical clindamycin 2 %, triamcinolone acetonide 0.1% solution
- Arm 3: Treat Only if Grade 3 Rash Occurs: Arm 3: Subjects (Approximately 50) that develop the rash caused by erlotinib will only be treated if their rash becomes severe to see if it will go away itself. The treatment for severe rash will be medicated lotion, (clindamycin 2% and hydrocortisone 1%,), applied to the rash and minocycline 100mg orally twice daily. Scalp lesions will be treated with a topical clindamycin 2 %, triamcinolone acetonide 0.1% solution
  clindamycin 2% and hydrocortisone 1%,: Arm 3: Subjects (Approximately 50) that develop the rash caused by erlotinib will only be treated if their rash becomes severe to see if it will go away itself. The treatment for severe rash will be medicated lotion, (clindamycin 2% and hydrocortisone 1%,), applied to the rash and minocycline 100mg orally twice daily. Scalp lesions will be treated with a topical clindamycin 2 %, triamcinolone acetonide 0.1% solution.
Arm/Group | Arm 1: Rash Prevention | Arm 2: Treat Only Upon Initiation of Rash | Arm 3: Treat Only if Grade 3 Rash Occurs
Serious Adverse Events (participants affected / at risk) | 1/49 | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 12/49 | 1/50 | 5/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Rash Prevention (N=49) | Arm 2: Treat Only Upon Initiation of Rash (N=50) | Arm 3: Treat Only if Grade 3 Rash Occurs (N=50)
Pancreatitis (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) — From treatment arm 1, however this SAE did not lead to discontinuation of treatment.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Rash Prevention (N=49) | Arm 2: Treat Only Upon Initiation of Rash (N=50) | Arm 3: Treat Only if Grade 3 Rash Occurs (N=50)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (General disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (General disorders) | 5 (5) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (2) | 0 (0) | 0 (0)
Decreased appetite (General disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (General disorders) | 2 (2) | 0 (0) | 2 (2)
Pancreatitis (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperbilirubinemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (General disorders) | 1 (1) | 0 (0) | 1 (1)
Headache (General disorders) | 0 (0) | 0 (0) | 1 (1)
Parsomia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Chromaturia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Dry Skin (General disorders) | 0 (0) | 1 (1) | 0 (0)
Skin Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Blister (General disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No